CLINICAL TRIAL: NCT00176748
Title: Phase 2 Study of the Anti-Angiogenesis Agent AG-013736 in Patients With Metastatic Thyroid Cancer Who Are Refractory to or Not Suitable Candidates for 131I Treatment
Brief Title: Treatment for Patients With Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Pfizer A4061014 - AG 013736 Study Katherine Liau, Pfizer, inc.and parexel, Int'l is the cro
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005-036; HUM 216
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AG 6013736

INTERVENTIONS:
Drug: AG 6013736 — 5 mg po bid

SUMMARY:
This study is being done to find out the good and bad effects of an investigational drug that is not approved for sale, called AG-013736. Tumors need blood vessels in order to continue to grow, and AG-013736 is thought to work by playing a role in preventing new blood vessels from growing. We want to see if AG-013736 has any effect on your disease by making your tumor smaller and if so, for how long. We also want to test the safety [the effect on your body] of AG-013736 and to measure the amount of AG-013736 that gets into your blood. AG-013736 has been given to over 140 patients with cancer on other studies.

DETAILED DESCRIPTION:
The American Cancer Society estimates that there will be about 23,600 new cases of thyroid cancer (5,960 in men and 17,640 in women) annually in the United States, and about 1,460 people (620 men and 840 women) will die from this disease.1 It is the most common malignancy of the endocrine system. Depending upon type and stage, thyroid cancer may be treated with surgery, radioactive iodine (131I), hormone treatment, external radiation, or chemotherapy.

The systemic therapy of metastatic disease remains palliative until new agents are found that might afford a better prognosis. Thyroid tumors are often vascular, and a decrease in the number of blood vessels that supply the tumor may starve it of needed nutrients. An approach to blocking the growth of blood vessels that supply the tumor is to inhibit the VEGF receptor tyrosine kinase (VEGFR TK) signaling pathway. The VEGFR TK inhibitor SU011248 has produced 4 objective responses in 15 patients receiving the drug on Phase 1 studies.2 AG-013736 is another VEGFR TK inhibitor. Besides having potential anti-angiogenesis properties through VEGFR TK inhibition, it also has additional potential antitumor through platelet derived growth factor receptor (PDGFR) TK inhibition.

ELIGIBILITY:
Inclusion Criteria

To be eligible for the study, subjects must satisfy all the following criteria:

1. Histologically documented thyroid cancer with metastases.
2. Failure of 131I to control the disease or 131I is not an appropriate therapy (eg, due to lack of iodine uptake by the tumor).
3. No expectation of further effects of prior anticancer therapy.
4. At least 1 target lesion, as defined by RECIST (Appendix C), that has not been irradiated. New lesions that have developed in a previously irradiated field may be used as sites of measurable disease assuming all other criteria are met. All target lesions must have a unidimensional diameter of at least 2 cm. (1 cm is acceptable for spiral CT scans if the reconstruction algorithm is 0.5 cm). Baseline measurements/evaluations must be completed within 4 weeks prior to treatment.
5. Adequate bone marrow, hepatic, and renal function documented within 14 days prior to treatment as documented by:

   * Absolute neutrophil count (ANC, calculated as the absolute number of neutrophils and bands) ≥1.5 x 109 cells/L
   * Platelets ≥100 x 109 cells /L
   * AST and ALT ≤2.5 x upper limit of normal (ULN), unless there are liver metastases in which case AST and ALT ≤5.0 x ULN
   * Total bilirubin ≤1.5 x ULN
   * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥60 mL/min
   * Urinary protein <2+ by urine dipstick. If dipstick is ≥2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours
6. Age ≥18 years.
7. ECOG performance status of 0 or 1 (see Appendix D)
8. No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be ≤140, and the baseline diastolic blood pressure readings must be ≤90. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
9. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to treatment.
10. Written and voluntary informed consent.

Exclusion Criteria

Subjects with one or more of the following criteria are ineligible for this study:

1. Central lung lesions involving major blood vessels (arteries or veins). (Central lesions that maintain the structural integrity of vessels have the potential to bleed if the tumor lesion undergoes necrosis. MRI or CT angiography should be used in any case where there is any question as to whether blood vessels are involved.)
2. History of hemoptysis
3. Gastrointestinal abnormalities including:

   * inability to take oral medication
   * requirement for intravenous alimentation
   * prior surgical procedures affecting absorption including gastric resection
   * treatment for active peptic ulcer disease in the past 6 months
   * active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy.
   * malabsorption syndromes.
4. Previous treatment with anti-angiogenesis agents including thalidomide, or inhibitors of epidermoid growth factor (EGF), platelet derived growth factor (PDGF), or fibroblast growth factors (FGF) receptors.
5. Current use or anticipated inability to avoid use of drugs that are known potent CYP3A4 inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, ergot derivatives, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, and delavirdine).
6. Current use or anticipated inability to avoid use of drugs that are known CYP3A4 or CYP1A2 inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, primidone, rifabutin, rifampin, and St. John's wort).
7. Active seizure disorder or evidence of brain metastases.
8. A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
9. History of a malignancy (other than thyroid cancer) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years
10. Major surgical procedure or any radiation therapy within 4 weeks of treatment.
11. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
12. Patients (male and female) having procreative potential who are not using adequate contraception or practicing abstinence
13. Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-07; Primary Completion 2006-08 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the response rate of AG-013736 in patients with metastatic thyroid cancer (who are refractory to or not suitable candidates for 131I treatment). | Approximately 2 years

SECONDARY OUTCOMES:
To determine the safety profile of AG-013736 | Approximately 2 years
To determine the progression-free survival | This is a variable in the outcome measure (time frame cannot be determined).
To determine the duration of response. | The time frame cannot be determined as it is the variable that is being studied for this Outcome Measure.
To determine overall survival. | Time Frame cannot be approximated as this is the variable that is being studied in this Outcome Measure.
To obtain blood samples for population pharmacokinetic analyses in order to explore relationships between clinical response and plasma soluble proteins. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis Worden, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States